CLINICAL TRIAL: NCT04554355
Title: Effects of a School-based Physical Activity Intervention for Fatness and Health-related Physical Fitness in Adolescents With Intellectual Disability
Brief Title: Effects of a PA Intervention for Fatness and Fitness in Adolescents With Intellectual Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, Gao Yang, Associate Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PHDSPE17482062
Record Dates: First submitted 2020-09-10; First posted 2020-09-18 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Obesity; Health-related Physical Fitness; Intellectual Disability
Keywords: Overweight; Obesity; Fitness; Adolescents; Intellectual disability
MeSH Terms: conditions — Obesity; Intellectual Disability; Overweight

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Outcomes Assessor
Masking Description: 1. those who entered data (student helpers) were exlcuded from fieldwork and intervention dilivery, data analysis and report writing.
  2. after data entry, only the PI knew the values of the two groups and stored the data separately in another file with passwords requested for access.
  3. data were analysed by a researcher, who was not involved in proposal writing and did not know which value means which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in this group will receive a three-month PA intervention (60 minutes/session, two sessions/week).
  Interventions: Behavioral: School-based PA intervention
- Control group (No Intervention): No intervention will be provided, participants in this group need to attend the regular school activities as normal.

INTERVENTIONS:
Behavioral: School-based PA intervention — Provide moderate to vigorous fun-game based exercises for adolescents with ID in schools to help them reduce obesity and improve fitness levels.
  Arms: Intervention group

SUMMARY:
The proposed study will be a 12-week school-based physical activity (PA) program with a 2-armed randomized controlled trial (RCT) design. It will target overweight and obese children with intellectual disability (ID). The primary outcomes will be both fatness-related and fitness-related outcomes. In addition, the effect of the intervention on blood pressure will be evaluated as the secondary outcomes.

DETAILED DESCRIPTION:
Childhood obesity and lower HRPF levels are major threats to public health. The previous research finds that children with ID are more vulnerable to be obesity and lower HRPF levels than general pediatric population. In addition, the transition from adolescence to young adulthood is recognized as a particularly high-risk period for weight gain. However, Interventions to reduce obesity and improve HRPF levels among adolescents with ID are scarce. The main purpose of this study is to implement and evaluate a fun game-based PA program to reduce overweight/obesity and improve health-related physical fitness (HRPF) levels among adolescents with ID (aged 12-18 years old).

The study consists of a 3-month intervention and a 3-month follow-up. Totally Forty-eight overweight/obese adolescents with mild intellectual disability (ID) will be recruited from special schools in China and then randomly assigned into two groups (n=24 for each group). Selection criteria for participants are: (1) children with mild ID; (2) aged 12-18 years old; (3) being overweight or obese; (4) without physical disability and other relevant health conditions. Participants in the experimental group will receive a fun game-based PA program (60 min/time, 2 sessions/week, 24 sessions totally) at school. No intervention will be provided to participants in the control group.

All participants in the two groups (N=48) will undertake repeated measurements on a set of study outcomes for three times. All measurements are non-invasive and no potential consequences are expected. In addition, questionnaires will be used to collect each participant's information of socio-demographic characteristics, physical activity level and eating habits (about 15 minutes).

The investigators expect the findings from the study would make up the knowledge gap and help eliminate existing health inequities among children with ID. It would serve as an example for use of other researchers, policy-makers, and the public to tackle off obesity among adolescents with ID in a global scale. If effective, this program would be welcomed and adopted by other special schools in the future. In addition, the effective model can also be extended to reach students with ID in normal schools.

ELIGIBILITY:
Inclusion Criteria:

* children with mild ID;
* aged 12-18 years old;
* overweight or obese;
* at least one family member who is able to attend the program with them.

Exclusion Criteria:

* with physical disability;
* with a medical predisposition towards obesity (such as genetic syndrome) that could interfere with the results of the study;
* with contraindications for PA (e.g. severe heart disease).

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Weight | up to 2 months
  It will be measured with a TANITA digital scale (TBF-410), which is accurate to 0.1 kg. The scale will be cleared before each participant is weighed, and the participants will be asked to remove any 'heavy' items from their pockets (keys, wallets etc.) and remove any heavy items of clothing or apparel (jackets, shoes, woollen jerseys etc.).
Weight | up to 5 months
  It will be measured with a TANITA digital scale (TBF-410), which is accurate to 0.1 kg. The scale will be cleared before each participant is weighed, and the participants will be asked to remove any 'heavy' items from their pockets (keys, wallets etc.) and remove any heavy items of clothing or apparel (jackets, shoes, woollen jerseys etc.).
Weight | up to 8 months
  It will be measured with a TANITA digital scale (TBF-410), which is accurate to 0.1 kg. The scale will be cleared before each participant is weighed, and the participants will be asked to remove any 'heavy' items from their pockets (keys, wallets etc.) and remove any heavy items of clothing or apparel (jackets, shoes, woollen jerseys etc.).
BMI | up to 2 months
  It will be calculated as weight (in kilograms) divided by the square of height (in metres) (kg/m2).
BMI | up to 5 months
  It will be calculated as weight (in kilograms) divided by the square of height (in metres) (kg/m2).
BMI | up to 8 months
  It will be calculated as weight (in kilograms) divided by the square of height (in metres) (kg/m2).
Waist circumference | up to 2 months
  It will be measured midway between the lowest rib margin and the top of the iliac crest at the end of a gentle expiration. The measure will be performed with a flexible metre ribbon accurate to 0.1 cm.
Waist circumference | up to 5 months
  It will be measured midway between the lowest rib margin and the top of the iliac crest at the end of a gentle expiration. The measure will be performed with a flexible metre ribbon accurate to 0.1 cm.
Waist circumference | up to 8 months
  It will be measured midway between the lowest rib margin and the top of the iliac crest at the end of a gentle expiration. The measure will be performed with a flexible metre ribbon accurate to 0.1 cm.
Hip circumference | up to 2 months
  It will be measured at the widest part of the body below the waist. The measurement of the waist circumference will be performed with a flexible metre ribbon accurate to 0.1 cm.
Hip circumference | up to 5 months
  It will be measured at the widest part of the body below the waist. The measurement of the waist circumference will be performed with a flexible metre ribbon accurate to 0.1 cm.
Hip circumference | up to 8 months
  It will be measured at the widest part of the body below the waist. The measurement of the waist circumference will be performed with a flexible metre ribbon accurate to 0.1 cm.
Waist to height ratio | up to 2 months
  The waist to height ratio will be calculated as waist circumference (in centimetres) divided by height (in centimetres).
Waist to height ratio | up to 5 months
  The waist to height ratio will be calculated as waist circumference (in centimetres) divided by height (in centimetres).
Waist to height ratio | up to 8 months
  The waist to height ratio will be calculated as waist circumference (in centimetres) divided by height (in centimetres).
Percent body fat | up to 2 months
  The percent body fat will be estimated with the TANITA digital scale (TBF-410) using foot-to-foot bioelectrical impedance analysis (BIA). After entering the participant's gender, race, height and age, the participant will be instructed to stand with bare feet on the metal footplates. The data will be displayed automatically.
Percent body fat | up to 5 months
  The percent body fat will be estimated with the TANITA digital scale (TBF-410) using foot-to-foot bioelectrical impedance analysis (BIA). After entering the participant's gender, race, height and age, the participant will be instructed to stand with bare feet on the metal footplates. The data will be displayed automatically.
Percent body fat | up to 8 months
  The percent body fat will be estimated with the TANITA digital scale (TBF-410) using foot-to-foot bioelectrical impedance analysis (BIA). After entering the participant's gender, race, height and age, the participant will be instructed to stand with bare feet on the metal footplates. The data will be displayed automatically.
6-min walk test | up to 2 months
  Testing procedures will follow Chow's study protocol (2018). The participants will be instructed and encouraged to cover the greatest possible distance on a flat surface 25 m in length. They will be instructed to keep a steady pace, whether running or walking. At the end of the test, the participants will be instructed to keep walking to aid in the recovery process. The distance will be measured by the number of laps around the track, adding extra distance as required (VOLEK et al., 2003). A trained examiner will measure and record the distance covered by each participant. Each participant will be assigned a trained partner (university student helper) based on his or her special physical condition and cognitive ability to give verbal direction and encouragement during the test.
6-min walk test | up to 5 months
  Testing procedures will follow Chow's study protocol (2018). The participants will be instructed and encouraged to cover the greatest possible distance on a flat surface 25 m in length. They will be instructed to keep a steady pace, whether running or walking. At the end of the test, the participants will be instructed to keep walking to aid in the recovery process. The distance will be measured by the number of laps around the track, adding extra distance as required (VOLEK et al., 2003). A trained examiner will measure and record the distance covered by each participant. Each participant will be assigned a trained partner (university student helper) based on his or her special physical condition and cognitive ability to give verbal direction and encouragement during the test.
6-min walk test | up to 8 months
  Testing procedures will follow Chow's study protocol (2018). The participants will be instructed and encouraged to cover the greatest possible distance on a flat surface 25 m in length. They will be instructed to keep a steady pace, whether running or walking. At the end of the test, the participants will be instructed to keep walking to aid in the recovery process. The distance will be measured by the number of laps around the track, adding extra distance as required (VOLEK et al., 2003). A trained examiner will measure and record the distance covered by each participant. Each participant will be assigned a trained partner (university student helper) based on his or her special physical condition and cognitive ability to give verbal direction and encouragement during the test.
30-second sit-to-stand | up to 2 months
  It will be used to assess participants' lower limb strength and endurance. It measures the maximum number of times a participant can rise to a full standing position from a seated position in a 30-second period, without pushing off with their arms. This test is administered using a school chair without arms, with a seat height around 14 inches (35.6 cm). The back of the chair will be placed against a wall to prevent it from moving. The participants will be instructed to sit in the middle of the chair, back straight, feet approximately shoulder width apart and placed on the floor at an angle slightly back from the knees, with one foot slightly in front of the other to help maintain balance. Arms are crossed at the wrists and held against the chest.
30-second sit-to-stand | up to 5 months
  It will be used to assess participants' lower limb strength and endurance. It measures the maximum number of times a participant can rise to a full standing position from a seated position in a 30-second period, without pushing off with their arms. This test is administered using a school chair without arms, with a seat height around 14 inches (35.6 cm). The back of the chair will be placed against a wall to prevent it from moving. The participants will be instructed to sit in the middle of the chair, back straight, feet approximately shoulder width apart and placed on the floor at an angle slightly back from the knees, with one foot slightly in front of the other to help maintain balance. Arms are crossed at the wrists and held against the chest.
30-second sit-to-stand | up to 8 months
  It will be used to assess participants' lower limb strength and endurance. It measures the maximum number of times a participant can rise to a full standing position from a seated position in a 30-second period, without pushing off with their arms. This test is administered using a school chair without arms, with a seat height around 14 inches (35.6 cm). The back of the chair will be placed against a wall to prevent it from moving. The participants will be instructed to sit in the middle of the chair, back straight, feet approximately shoulder width apart and placed on the floor at an angle slightly back from the knees, with one foot slightly in front of the other to help maintain balance. Arms are crossed at the wrists and held against the chest.
One minute sit-up | up to 2 months
  will be adopted to evaluate participants' abdominal muscular strength and endurance. The task is to perform as many sit-ups as possible in one minute, or until the participant experiences muscle fatigue and cannot try any more. The participants will be instructed to cross their arms on their chests with hands on shoulders, and to tighten their abdominal muscles and rise up to touch elbows to thighs. Then, they return to the start position and repeat.
One minute sit-up | up to 5 months
  will be adopted to evaluate participants' abdominal muscular strength and endurance. The task is to perform as many sit-ups as possible in one minute, or until the participant experiences muscle fatigue and cannot try any more. The participants will be instructed to cross their arms on their chests with hands on shoulders, and to tighten their abdominal muscles and rise up to touch elbows to thighs. Then, they return to the start position and repeat.
One minute sit-up | up to 8 months
  will be adopted to evaluate participants' abdominal muscular strength and endurance. The task is to perform as many sit-ups as possible in one minute, or until the participant experiences muscle fatigue and cannot try any more. The participants will be instructed to cross their arms on their chests with hands on shoulders, and to tighten their abdominal muscles and rise up to touch elbows to thighs. Then, they return to the start position and repeat.
Handgrip strength | up to 2 months
  It will be used to assess participants' hand and forearm muscular strength. During the test, the participant will be instructed to adopt a standing position, with arms at his/her side, not touching the body. The participant will be asked to squeeze the dynamometer with as much force as possible, being careful to squeeze only once for each measurement. Three trials will be made with a pause of 10-20 s between each to avoid the effects of muscular fatigue. Right and left hands will be alternated. The best score will be recorded.
Handgrip strength | up to 5 months
  It will be used to assess participants' hand and forearm muscular strength. During the test, the participant will be instructed to adopt a standing position, with arms at his/her side, not touching the body. The participant will be asked to squeeze the dynamometer with as much force as possible, being careful to squeeze only once for each measurement. Three trials will be made with a pause of 10-20 s between each to avoid the effects of muscular fatigue. Right and left hands will be alternated. The best score will be recorded.
Handgrip strength | up to 8 months
  It will be used to assess participants' hand and forearm muscular strength. During the test, the participant will be instructed to adopt a standing position, with arms at his/her side, not touching the body. The participant will be asked to squeeze the dynamometer with as much force as possible, being careful to squeeze only once for each measurement. Three trials will be made with a pause of 10-20 s between each to avoid the effects of muscular fatigue. Right and left hands will be alternated. The best score will be recorded.
Sit to reach test | up to 2 months
  Each participant will begin the test by removing his/her shoes (very thin footwear will be permitted) and sitting down at the test apparatus. One leg will be fully extended with the foot flat against the end of the testing instrument. The other knee will be bent, with the sole of the foot flat on the floor 5-8 cm to the side of the straight knee. The arms will be extended forward over the measuring scale with hands palms down, one on top of the other. Each participant will be instructed to reach directly forward with both hands along the scale four times and to hold the position of the fourth reach for at least 1 s. After measuring one side, the participant will be asked to switch the position of his/her legs and reach again. The participant can allow the bent knee to move to the side if necessary as the body moves forward.
Sit to reach test | up to 5 months
  Each participant will begin the test by removing his/her shoes (very thin footwear will be permitted) and sitting down at the test apparatus. One leg will be fully extended with the foot flat against the end of the testing instrument. The other knee will be bent, with the sole of the foot flat on the floor 5-8 cm to the side of the straight knee. The arms will be extended forward over the measuring scale with hands palms down, one on top of the other. Each participant will be instructed to reach directly forward with both hands along the scale four times and to hold the position of the fourth reach for at least 1 s. After measuring one side, the participant will be asked to switch the position of his/her legs and reach again. The participant can allow the bent knee to move to the side if necessary as the body moves forward.
Sit to reach test | up to 8 months
  Each participant will begin the test by removing his/her shoes (very thin footwear will be permitted) and sitting down at the test apparatus. One leg will be fully extended with the foot flat against the end of the testing instrument. The other knee will be bent, with the sole of the foot flat on the floor 5-8 cm to the side of the straight knee. The arms will be extended forward over the measuring scale with hands palms down, one on top of the other. Each participant will be instructed to reach directly forward with both hands along the scale four times and to hold the position of the fourth reach for at least 1 s. After measuring one side, the participant will be asked to switch the position of his/her legs and reach again. The participant can allow the bent knee to move to the side if necessary as the body moves forward.

SECONDARY OUTCOMES:
Blood pressure (both diastolic and systolic blood pressure) | up to 2 months
  It will be measured using an Omron blood pressure monitor. (It will be calibrated before using.) During the test, the participant will be asked to sit quietly for about 5 minutes, and then to remove outer garments and roll up their shirt sleeves if necessary to bare the upper right arm. The measurements will be taken on the right arm whenever possible. The participant's arm will be resting on the desk so that the antecubital fossa is at the level of the heart and with the palm relaxed and facing upwards. Then, the cuff will be placed on the right arm, with the bottom edge 1-2 cm above the antecubital fossa. The top edge of the cuff cannot be restricted by clothing.
Blood pressure (both diastolic and systolic blood pressure) | up to 5 months
  It will be measured using an Omron blood pressure monitor. (It will be calibrated before using.) During the test, the participant will be asked to sit quietly for about 5 minutes, and then to remove outer garments and roll up their shirt sleeves if necessary to bare the upper right arm. The measurements will be taken on the right arm whenever possible. The participant's arm will be resting on the desk so that the antecubital fossa is at the level of the heart and with the palm relaxed and facing upwards. Then, the cuff will be placed on the right arm, with the bottom edge 1-2 cm above the antecubital fossa. The top edge of the cuff cannot be restricted by clothing.
Blood pressure (both diastolic and systolic blood pressure) | up to 8 months
  It will be measured using an Omron blood pressure monitor. (It will be calibrated before using.) During the test, the participant will be asked to sit quietly for about 5 minutes, and then to remove outer garments and roll up their shirt sleeves if necessary to bare the upper right arm. The measurements will be taken on the right arm whenever possible. The participant's arm will be resting on the desk so that the antecubital fossa is at the level of the heart and with the palm relaxed and facing upwards. Then, the cuff will be placed on the right arm, with the bottom edge 1-2 cm above the antecubital fossa. The top edge of the cuff cannot be restricted by clothing.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Gao, PhD, Principal Investigator — Hong Kong Baptist University; Aiwei Wang, Master, Study Director — Hong Kong Baptist University
Locations (1):
- Hong Kong Bapist University, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang A, Bu D, Yu S, Sun Y, Wang J, Lee TCT, Baker JS, Gao Y. Effects of a School-Based Physical Activity Intervention for Obesity, Health-Related Physical Fitness, and Blood Pressure in Children with Intellectual Disability: A Randomized Controlled Trial. Int J Environ Res Public Health. 2022 Sep 22;19(19):12015. doi: 10.3390/ijerph191912015. PMID 36231316
- [Derived] Wang A, Gao Y, Wang J, Tong TK, Sun Y, Yu S, Zhao H, Zou D, Zhang Z, Qi Y, Zuo N, Bu D, Zhang D, Xie Y, Baker JS. Effects of a School-Based Physical Activity Intervention for Obesity and Health-Related Physical Fitness in Adolescents With Intellectual Disability: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Mar 22;10(3):e25838. doi: 10.2196/25838. PMID 33749611